CLINICAL TRIAL: NCT00519194
Title: CONcomitant eValuation of Epicor Left atRial Therapy for AF
Acronym: CONVERT-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 051.13
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: Arrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epicor Cardiac Ablation (Experimental)
  Interventions: Device: Epicor LP Cardiac Ablation System; Procedure: Surgical ablation of permanent AF

INTERVENTIONS:
Device: Epicor LP Cardiac Ablation System — Surgical ablation of permanent AF during concomitant open chest and/or open heart surgery
Procedure: Surgical ablation of permanent AF — Concomitant AF ablation during mitral valve surgery

SUMMARY:
The purpose of this study is to test the safety and efficacy of the Epicor LP Cardiac Ablation System for treating permanent atrial fibrillation during concomitant open chest and/or open heart surgery for one of more of the following procedures: mitral valve repair or replacement, aortic valve repair or replacement, tricuspid valve repair or replacement, coronary artery bypass surgery or patent foramen ovale (PFO closure).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Permanent AF defined as continuous AF lasting > one year OR non self-terminating AF lasting > seven days but no more than one year with at least one failed DC cardioversion
* Have a concomitant indication for open chest and/or open heart surgery for one or more of the following: mitral valve repair or replacement, aortic valve repair or replacement, tricuspid valve repair or replacement, patent foramen ovale (PFO) closure or coronary artery bypass surgery
* Be able to take anticoagulation therapy
* Be able to fulfill study requirements
* Be able to sign study-specific informed consent

Exclusion Criteria:

* Presence of a previously implanted device in or adjacent to the treatment target area that may alter the delivery of therapy
* Prior cardiac surgery
* Presence of active endocarditis, local or system infection
* Presence of advanced heart failure (NYHA class > II, & LVEF < 20%)
* Intraaortic balloon pump, IV inotropes or vasoactive agents within 30 days
* Emergent cardiac surgery due to acute MI or acute mitral regurgitation
* Life expectancy < 1 year
* Major or progressive non-cardiac disease
* Presence of left atrial thrombi
* Left atrial diameter > 6.0 cm
* Any condition that prevents investigator from safely performing procedure
* Positive urine or serum pregnancy test
* Prior left atrial ablation
* Currently participating in another clinical research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Groh, MD, Principal Investigator — Mission Hospitals
Locations (15):
- United States (15):
  - St. Agnes Medical Center, Fresno, California
  - Manatee Memorial Hospital, Bradenton, Florida
  - Blake Medical Center, Bradenton, Florida
  - Cardiology Consultants, MD's PA (Baptist Hospital), Pensacola, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Community Hospital, Munster, Indiana
  - Midatlanatic Cardiovascular Associates, PA; Union Memorial Hospital, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation/Abbott NW Hospital, Minneapolis, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Mission Hospital, Inc, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Epicor Cardiac Ablation: Epicor LP Cardiac Ablation System: Surgical ablation of permanent AF during concomitant open chest and/or open heart surgery
  Surgical ablation of permanent AF: Concomitant AF ablation during mitral,aortic, and or tricuspid valve surgery, PFO closure or CABG procedure
Period: Overall Study
Arm/Group | Epicor Cardiac Ablation
Started | 112
Completed | 91
Not Completed | 21
Not completed — Withdrawal by Subject | 9
Not completed — Death | 9
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Subjects treated
Arm/Group | Epicor Cardiac Ablation
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 67
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Atrial Fibrillation in the Absence of Any AF Therapies
Description: Freedom from atrial fibrillation (AF) at 6 months in absence of any AF therapies.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Epicor Cardiac Ablation
Number analyzed (Participants) | 91
participants | 49

ADVERSE EVENTS:
Arm/Group | Epicor Cardiac Ablation
Serious Adverse Events (participants affected / at risk) | 11/112
Other Adverse Events (participants affected / at risk) | 1/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epicor Cardiac Ablation (N=112)
Cardiac injury related to Epicor device rsulting in unplanned surgical or catheter intervention (Cardiac disorders) | 1 (1)
Death (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Newly developed third degree AV block requiring permanent pacemaker implantation (Cardiac disorders) | 4 (4)
Peripheral arterial embolism (Vascular disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epicor Cardiac Ablation (N=112)
Acute heart failure (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No